CLINICAL TRIAL: NCT06073548
Title: Patient Experience and Quality of Life During the Surveillance Phase of Uveal Melanoma: A Prospective Multi-method Study
Acronym: SALOME Quali
Status: Not yet recruiting | Type: Observational
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: IC 2022-11
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Uveal Melanoma
Keywords: Uveal Melanoma; Ophtalmic oncology; Quality of life; Fear of recurrence; Communication
MeSH Terms: conditions — Uveal Melanoma; Communication | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires and interviews — Patients wiill be asked to fulfill questionnaires at inclusion and 6 months after. An interview will be offered to a sub-sample of patients (approximately 20 patients).

SUMMARY:
The goal of this prospective observational study is to learn about patient quality of life and experience and medical information needs during uveal melanoma post-treatment surveillance. Participants have previously undergone treatment for non-metastatic uveal melanoma and have integrated a oncological and / or ophthalmic surveillance protocol based on their individual genomic and / or clinical risk of recurrence. The main objectives it aims to assess are:

* To evaluate the effect of satisfaction with communication with the oncologist/ophthalmologist during the oncology/ophthalmology surveillance visit 6 months after the start of surveillance (T1) on the overall level of health status/quality of life (QoL).
* To explore the impact on psychosocial resources and needs such as fear of recurrence, anxiety and depression 6 months after the start of surveillance (T1) and 12 months after the start of surveillance (T2).
* To document patients experience of care and communication during the first 12 months of surveillance.

Participants will fill in quality of life questionnaires at two timepoints. A sub-sample will be offered to participate in qualitative research interviews. Researchers will compare data from patients at low risk of recurrence with those at high risk of recurrence to see if there are significant differences with regards to quality of life, satisfaction with care and medical information needs.

DETAILED DESCRIPTION:
Context and scientific background Uveal melanoma (UM) is the most common malignant ocular tumour in adults. It is a rare disease with an incidence of four to seven new cases per million per year in western countries (Mathis, 2018). The diagnosis of uveal melanoma is usually made when vision problems appear and the disease is still at a localized stage (in 95% of cases). Historically, the standard treatment for uveal melanoma was enucleation. Today, around 75% of patients can benefit from conservative treatment approaches such as brachytherapy or proton beam therapy without increasing the risk of metastasis or affecting survival. The visual prognosis of uveal melanoma depends on the localization of the tumour and efficacy of the treatment. Vital prognosis depends on the metastatic risk, which is related to the tumours' size and genomic characteristics (AJCC 7th Edition, 2015).

Up to 50% of patients develop metastases within a median time range of 2 to 3 years (Tuomaala & Kivelä, 2004). Metastatic progression develops most frequently in the liver (in >80% of cases). Once the disease spreads to the liver, median survival ranges from 3 to 12 months (Mariani, 2012) and response to treatment is rare. Estimating metastatic risk allows to provide personalized surveillance. For high risk patients, current international recommendations (NICE 2015) advise surveillance with liver CT or MRI (magnetic resonance imaging) every 6 months for over 10 years. If uveal melanoma metastases are diagnosed early, surgical liver resection can be considered in 25% of patients (Mariani, 2016). For the remaining 75%, systemic palliative care is recommended.

Various studies have addressed the effects of localized uveal melanoma and its treatment on quality of life (QoL). The QoL of patients with uveal melanoma appears to be significantly lower compared to matched general population (Erim, 2016; Miniati, 2018). Within the two years after treatment, overall QoL appears to be similar in patients treated by either enucleation or radiotherapy (Hope-Stone, 2016). Furthermore, no difference has been found between these treatments regarding specific aspects of QoL such as the ability to drive, ocular irritation, headaches, concerns regarding body image, and fear of recurrence (Hope-Stone, 2019). However, 6 months after treatment, functional difficulties are more important in enucleated patients, whereas difficulties in central and peripheral vision as well as in reading are higher in patients treated by radiotherapy (Hope-Stone, 2019). A large prospective study, conducted over a 20 year-period, concluded that overall quality of life was worse in enucleated patients than in patients treated with radiotherapy. However, this difference is not attributed to the treatment but to factors predisposing to treatment choices such as a more severe disease (e.g., larger tumour) (Damato, 2018).

During post-treatment surveillance, important aspects of QoL appear to be altered in patients treated for uveal melanoma. Depression and QoL levels seem to be worse around three months post-treatment (Amaro, 2010). Specific problems affecting QoL persist such such as body image troubles, especially in enucleated patients, as well as psychological adjustment, and social functioning difficulties, especially when vision problems persist.

As reported by items of the EORTC QLQ-C30 questionnaire, 39% of patients may have significant vision problems and 33% may report being 'worried about their future health' (Frenkel, 2018). The latter issue refers to fear of cancer recurrence (FCR) which is defined as the "fear, worry, or concern relating to the possibility that cancer will come back or progress" (Lebel, 2016). It is characterized by intense worry, intrusive thoughts and difficulty planning the future. Fear of recurrence (Suchocka-Capuano, 2011; Damato, 2018) has shown to be high and persists over time. These fears are related to uncertainty regarding future health. They result in anxiety and depressive symptoms, which significantly affect overall quality (Hope-Stone, 2015). Risk factors predisposing to distress include tumour stage and time since the beginning of surveillance. (Klingenstein, 2020) and persistent or emerging post-treatment symptoms and functional limitations (Brown, 2021). To our knowledge, only one study has examined unmet needs in patients with non-metastatic uveal melanoma, highlighting significant unmet medical information and psychological needs within 1 week after diagnosis and 3 months later (Williamson, 2018).

Prognostication tools based on clinical and genomic factors are available in routine practice (Cassoux, 2014). These tools may be used in consultation to inform cancer patients about the estimated risk of recurrence and associated life expectancy. Studies evaluating the psychosocial impact of communicating genomic test results and informing patients about their risk of cancer recurrence have been conducted primarily with breast cancer patients to guide the choice of adjuvant therapy. They suggest that a poor understanding of genomic tests results leads to increased anxiety (Pellegrini, 2012). Higher levels of anxiety are also related to lower satisfaction with having this testing done (Tzeng, 2010). Regarding the utilization of these tests in patients with uveal melanoma, studies from Anglo-Saxon countries report that many patients want to be informed of the genomic test result indicating their risk of metastatic recurrence (Beran, 2009; Damato, 2013; Brown, 2020). Risk estimations are provided in the form of numbers accompanied by graphs or pictograms to help interpret and understand the information, and thus enable informed decision-making concerning care and monitoring. However, a significant number of patients also experience regrets about being informed of their genomic test result and risk of recurrence, regardless of their personal risk status (Schuermeyer, 2016).

MRI appears to be the most sensitive screening method available for the early detection of metastases (Piperno-Neumann, 2015). Institut Curie has developed a clinical trial in which patient surveillance is tailored based on the risk of metastatic recurrence. In this trial, patients at high risk of recurrence receive liver MRI every 6 months. As for patients at high risk intense surveillance in terms of frequency and type of medical testing is recommended, patients may know that they have a higher risk of disease recurrence. However, there is no scientific data on this. Therefore, it is important to assess how patients with uveal melanoma at high risk of recurrence perceive the information provided by the oncologist (e.g. regarding risk of recurrence testing) and to evaluate its impact on quality of life, and more precisely, fear of recurrence. In general, cancer patients whose information needs are met have better QoL and lower levels of anxiety and depression (Husson, 2011). Nevertheless, up to now, we have little knowledge about the relation between information needs and QoL in UM patients (Lieb, 2020). This study shows that prognostic testing may help to alleviate distress and promote more realistic risk perception. Furthermore, even less information exists in French culture, where the communication of precise numeric estimations of recurrence risk may not be well accepted. Cultural factors affect patients' care needs, their expectations and expression of wishes, and influence clinicians' attitude in the relationship and communication with patients. Specifically, Anglo-Saxon cultures tend to value self-determination and autonomy, which impact the amount, precision and timing process of the medical information requested or provided in situations of medical uncertainty (Razavi, 2019).

Moreover, most studies on quality of life and psychosocial needs in patients affected with UM as cited above are conducted in countries with an Anglo-Saxon culture (Schuermeyer, 2016; Damato, 2018; Hope-Stone, 2019). Studies performed in other countries do not have a prospective design (Moschos, 2018; Frenkel, 2018) and use heterogeneous quality of life assessments which make comparisons and synthesis of results difficult (Miniati, 2018). To sum up, we lack robust, prospective data on needs and satisfaction with type and amount of information provided and their impact on QoL in French cancer patients with either a confirmed high risk or low risk of relapse. Advances in prognostication of cancer recurrence and identification of predictive biomarkers of response to treatment in oncology as well as the availability of genomic tests in clinical practice (Cassoux, 2014; Piperno-Neumann, 2019), increase the importance to evaluate how French patients perceive medical communication about the results of these tests and their impact on QoL and fear of metastatic relapse.

A patient-centered approach seems to enhance QoL (Brédart, 2013; Castro, 2016). Patient-centered care entails attention to the patient's communication needs, personalized information, emotional support, care coordination and continuity. This kind of approach promotes patient's ability to remember medical information, understanding of medical recommendations, and satisfaction with care. Furthermore, it can minimize uncertainty and distress. In the context of uveal melanoma, patients may expect information regarding their risk of metastatic recurrence, which enables them to anticipate potential medical and/or personal consequences (e.g., on medical follow-up, personal life choices). In this context, some patients may need major attention and emotional support from their physician. A referral to psychological counselling and further supportive care may also be helpful (Hope-Stone, 2018).

In uveal melanoma, the information of high metastatic recurrence risk is generally communicated by an oncologist to whom the patient is referred and who implement a first oncology surveillance visit (~ 2 months post-treatment). This patient generally does not see his/her hospital ophthalmologist anymore. In contrast, UM patients at low risk of recurrence continue to be follow-up by this specialist in collaboration with an extra-hospital ophthalmologist. Patients' QoL and fear of recurrence may be affected by their satisfaction with the interactions with clinicians and cancer care services. For UM patients these aspects are thus relevant in terms of patient-reported outcomes. Studies with breast cancer patients have shown that sharing emotions with physicians can reduce fear of recurrence after radiation therapy. It reflects the effect of communication processes on this aspect of QoL (Humphris, 2019). To our knowledge, the association between the patients' satisfaction with information and their QoL and fear of recurrence has never been explored in the context of non-metastatic uveal melanoma at either high or low recurrence risk.

Methodology This is a single-centre, prospective observational study, which combines a quantitative and qualitative research approach. This mixed method design will enable to explore the relationships between patients' experience of communication with the oncologist, and quality of life, and fear of recurrence.

At six months (+/- one month) after the end of treatment (T1), patients will be invited to participate in the study. They will be invited to complete a set of questionnaires, including the EORTC QLQ-C30, EORTC QLQ-OPT30 quality of life questionnaires and the FCRI Fear of cancer recurrence inventory. Patients will be invited to complete some of these measures again at T2, i.e. 12 months (+/- one month) post-treatment. Clinical data will be collected at T1 by the researcher.

A complementary sequential qualitative study will be conducted involving a random sub-sample of the study population after completion of questionnaires. A purposive sampling will target an equivalent number of patients per UM treatment (enucleation vs radiotherapy only) and surveillance modality (MRI for high risk vs CT scan only for low risk).

An interview guide will be developed to explore: how oncologist- or ophthalmologist-patient interactions potentially relate to fear of recurrence and quality of life during the first 6-month of follow-up; how oncologist or ophthalmologist-patient interactions can minimize the effect of factors such as physical symptoms and functional limitations which are likely risk factors for persistent fear of recurrence (Brown, 2021); what about the more intensive follow-up of uveal melanoma at high risk of recurrence, the information given and their impact on fear of recurrence and quality of life? Data are collected using psychometrically validated questionnaires, items adapted from the literature and from the medical records for age, gender and clinical information.

The EORTC QLQ-C30 (30 items) (Aaronson, 1993) is used to assess functioning difficulties, symptoms and general aspects of quality of life.

The EORTC QLQ-OPT30 module (30 items) (Brandberg, 2004) will be used to measure aspects of quality of life specific to ocular cancers and their treatments (e.g., ocular irritation or difficulties with daily activities).

For both the QLQ-C30 and QLQ-OPT30, a score from one to 100 is calculated on each scale. A high score for a functional scale or the global health status/QoL denotes high/healthy level of functioning and high QoL, while high score on symptom scales denotes high level of symptomatology/problem.

The FCRI (42 items) (Simard, 2009) measures fear of cancer recurrence in seven factors: Triggers, Severity, Psychological Distress, Coping Strategies, Functioning impairments, Insight, and Reassurance. The total score ranges from 0 to 168. A higher score indicates a higher level of fear of recurrence. A cut-off score of 13 on the FCRI Severity Subscale was found to be associated with optimal sensitivity and specificity for detection of clinical levels of FCR.

Anxiety and depression are assessed by the HADS (14 items) (Zigmond & Snaith, 1983; VF Razavi et al., 1990). This questionnaire includes 14 items whose answers are scored 0 to 3 Higher scores indicate higher levels of anxiety and/or depression.

The EORTC QLQ-INFO25 (25 items) (Arraras et al., 2010) is used to assess the perception of information about the disease and treatment. It is composed of 4 multi-item scales (information about disease, medical tests, treatment and other services) and eight single items. Response to each item are scored from 1 to 4. The sum of scores by dimension is transformed into a score from 0 to 100 scale. A high score on a given subscale indicates a higher amount of received information or of higher levels of satisfaction. Among single items, one addresses the wish to receive additional information and another the wish to receive less information, with response options yes versus no.

Multi-item subscales of the EORTC PATSAT-C33 (27 items) (Brédart, 2018) are used to assess technical skills, information exchange and interactions with physicians; and services and organisation of care in terms of coordination of care and interactions with all care professionals. In this project we will also use a single item assessing overall quality of care.

The multi-item scales or single items are scored in a similar way: (1) the scores of the individual items in a scale are first summed up and then, for multi-item scales, divided by the number of items in the scale; (2) these single item/scale scores are then transformed in order to obtain a score range from 0 to 100, with a higher score representing a higher level of satisfaction with care/perceived quality of care.

Data collected from clinicians: Perception of the surveillance consultation as well as satisfaction with the consultation are assessed by a 6-items questionnaire similar to the questionnaire addressed to patients.

ELIGIBILITY:
* Patient aged 18 years or older.
* Diagnosed with a non-metastatic uveal melanoma
* Completion of primary tumour treatment ≥ 6 months (+/- two months).
* Able to respect scheduled visits.
* Able to read and understand the language of the questionnaires.

Two groups of patients will be identified:

1. Patients with non-metastatic uveal melanoma at high risk for metastatic relapse defined as:

   * T2b/c/d or ≥ T3,
   * or anomaly on either chromosome 3 or chromosome 8, found by CGH array or sequencing.
2. Patients with non-metastatic uveal melanoma at low risk of recurrence defined as:

   * T2a,

     * and/or no alteration of chromosome 3 or chromosome 8 has been found.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Newly patients undergoing surveillance for non-metastatic UM will be consecutively included either at the oncologist (for high-risk patients) or ophthalmologist (for low risk patients) consultation. Those at high risk of metastatic recurrence are those taking part of a cohort including 700 patients with non-metastatic uveal melanoma at high risk of metastatic recurrence, whose aim is to provide intensive clinical surveillance (MRI every 6 months) based on risk of UM metastatic recurrence. Patients at low risk of metastatic recurrence are followed by the ophthalmologist and receive liver ultrasound every 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of satisfaction with communication with the oncologist/ophthalmologist during the oncology/ophthalmology surveillance visit on the overall level of health status/quality of life (QoL). | At T1, 6 months after the start of surveillance.
  EORTC QLQ-INFO25 item on overall satisfaction with information

SECONDARY OUTCOMES:
To document the experience of surveillance consultations for uveal melanoma patients at high risk of recurrence versus low risk of recurrence, from the point of view of patients and clinicians. | At T1, 6 months after the start of surveillance.
  Communication experience will be assessed by analogue patient and clinician questions (perception of information and communication, knowledge related to examinations and prognostic testing, benefits and risks of providing medical information, particularly concerning the risk of metastatic recurrence). Furthermore, clinicians years of experience will be assessed.
To document the satisfaction of patients at high and low risk of metastatic recurrence with organization of the surveillance phase (e.g. coordination, continuity of care). | At T1 (i.e. 6 months from the start of the surveillance phase).
  Subscale coordination of the EORTC PATSAT-C33 module will be used to compare level of satisfaction in patient at high versus low risk of recurrence.
To evaluate the effect of satisfaction of patients at high versus low risk of recurrence with regard to communication with the oncologist / ophthalmologist on fear of recurrence. | At T1 and then at T2 (i.e. at six and 12 months from the start of the surveillance phase).
  The subscale "doctors" of the EORTC PATSAT-C33 will assess satisfaction with care and satisfaction with communication will be assessed by the EORTC QLQ-INFO25, at T1 each. Their effect on Fear of cancer recurrence will be measured by the FCRI at T1 and T2.
To explore coping strategies and preferences with regard to medical information, particularly concerning medical examinations and prognostic tests, in patients at high and low risk of metastatic recurrence. | At T1 (i.e. 6 months from the start of the surveillance phase).
  Coping strategies will be assessed by the subscale of FCRI.
To identify the psycho-social needs and assess the quality of life (e.g. anxiety, depression) of patients at high and low risk of metastatic recurrence, as well as changes in these needs over time. | At inclusion and then at T2 (i.e. 6 and 12 months respectively from the start of the oncological surveillance phase).
  Different dimensions of quality of life will be assessed by the EORTC QLQ-C30. Anxiety and depression will be measured with HADS, furthermore additional items will assess the wish for psychological counselling. EORTC QLQ-OPT30 will assess symptoms and how the modulate quality of life and especially psychosocial variables.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Muller A, Dolbeault S, Piperno-Neumann S, Clerc M, Jarry P, Cassoux N, Lumbroso-Le Rouic L, Matet A, Rodrigues M, Holzner B, Malaise D, Bredart A. Anxiety, depression and fear of cancer recurrence in uveal melanoma survivors and ophthalmologist/oncologist communication during survivorship in France - protocol of a prospective observational mixed-method study. BMC Psychiatry. 2024 Nov 15;24(1):812. doi: 10.1186/s12888-024-06265-2. PMID 39548476